CLINICAL TRIAL: NCT01735214
Title: An Observational Study of Patients With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT) Who Switched IOP-lowering Treatments
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/GLA/037
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Results first posted 2015-04-27 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with POAG or OHT: Patients with POAG or OHT on current IOP-lowering therapy who are prescribed a prostaglandin analogue -containing IOP-lowering therapy by the physician. The decision to prescribe a change in IOP-lowering therapy lies with the physician according to their standard practice.
  Interventions: Drug: Prostaglandin Analogue -Containing IOP-Lowering Therapy

INTERVENTIONS:
Drug: Prostaglandin Analogue -Containing IOP-Lowering Therapy — Patients with POAG or OHT on current IOP-lowering therapy who are prescribed a prostaglandin analogue -containing IOP-lowering therapy by the physician. The decision to prescribe a change in IOP-lowering therapy lies with the physician according to their standard practice.

SUMMARY:
This study is a prospective, observational study of changing from any IOP-lowering treatment to a prostaglandin analogue-containing IOP-lowering medication for patients with Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT). The decision to change medications lies with the physician according to their standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open angle glaucoma (POAG) or ocular hypertension (OHT)
* Previously prescribed any IOP-lowering therapy which has been stopped and a new prostaglandin analogue -containing IOP-lowering therapy started

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: POAG or OHT
Sampling Method: Non-Probability Sample
Enrollment: 358 (Actual)
Dates: Start 2013-03-07 (Actual); Primary Completion 2014-04-10 (Actual); Study Completion 2014-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Tamcelik N, Izgi B, Temel A, Yildirim N, Okka M, Ozcan A, Yuksel N, Elgin U, Altan C, Ozer B. Prospective, non-interventional, multicenter study of the intraocular pressure-lowering effects of prostaglandin analog/prostamide-containing therapies in previously treated patients with open-angle glaucoma or ocular hypertension. Clin Ophthalmol. 2017 Apr 19;11:723-731. doi: 10.2147/OPTH.S119963. eCollection 2017. PMID 28458511

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With POAG or OHT
Started | 358
Completed | 358
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 358
Age, Customized [Number; unit: participants]
  18 to 30 years | 10
  31 to 40 years | 9
  41 to 50 years | 28
  51 to 60 years | 89
  61 to 70 years | 125
  71 to 80 years | 81
  81 to 90 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 178

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) in the Right Eye
Description: IOP is a measurement of the fluid pressure inside the eye. A negative change from Baseline indicates an improvement.
Time Frame: Baseline, Week 12
Population: All participant with IOP data at Baseline and Week 12 for analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 312
mmHg | -4.5 (4.6)

2. Secondary Outcome: Patient Assessment of Overall Tolerability With New Treatment Using a 4-Point Scale
Description: The patient evaluated the tolerability of IOP-lowering medication therapy using a 4-Point Scale: Very good, Good, Moderate or Poor. Percentage of participants in each category is reported.
Time Frame: 12 Weeks
Population: All participants with available data.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 358
percentage of participants
  Very good | 48.6
  Good | 31.6
  Moderate | 6.1
  Poor | 1.7
  Missing data | 12.0

3. Secondary Outcome: Physician Assessment of Tolerability With New Treatment Using a 4-Point Scale
Description: The physician evaluated the patient's tolerability of IOP-lowering medication therapy using a 4-Point Scale: Very good, Good, Moderate or Poor. Percentage of participants in each category is reported.
Time Frame: 12 Weeks
Population: All participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 358
percentage of participants
  Very good | 50.0
  Good | 33.0
  Moderate | 4.7
  Poor | 2.2
  Missing data | 10.1

4. Secondary Outcome: Percentage of Participants Who Discontinue the Use of New Treatment Prior to 12 Weeks
Time Frame: 12 Weeks
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 358
percentage of participants | 7.5

5. Secondary Outcome: Percentage of Participants Who Continue the New Treatment After 12 Weeks
Time Frame: 12 Weeks
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 358
percentage of participants | 83.5

6. Secondary Outcome: Physician Assessment of Adherence to New Treatment Using a 4-Point Scale
Description: The physician assessed the participant's adherence to new treatment using the following scale: Not Applicable, Worse, Equal or Better. The percentage of participants in each category is reported.
Time Frame: 12 Weeks
Population: All Participants
Measure: Number; unit: percentage of participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 358
percentage of participants
  Not Applicable | 1.68
  Worse | 4.47
  Equal | 42.74
  Better | 41.34
  Missing data | 9.78

7. Secondary Outcome: Physician Assessment of Efficacy Using a 5-Point Scale
Description: The physician evaluated efficacy (IOP lowering) using a 5-Point Scale: IOP lower than target, Reached Target IOP, IOP decreased but target not reached, No change or IOP increased. The percentage of participants in each category is reported.
Time Frame: 12 Weeks
Population: All participants.
Measure: Number; unit: percentage of participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 358
percentage of participants
  IOP lower than target | 24.0
  Reached target IOP | 49.7
  IOP decreased but target NOT reached | 10.9
  No change | 0.8
  IOP increased | 4.7
  Missing data | 9.8

8. Secondary Outcome: Percentage of Participants Reaching Individual IOP Target After 12 Weeks
Time Frame: 12 Weeks
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 358
percentage of participants | 49.7

9. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) in the Left Eye
Description: IOP is a measurement of the fluid pressure inside the eye. A negative change from Baseline indicates an improvement.
Time Frame: Baseline, Week 12
Population: All participant with IOP data at Baseline and Week 12 for analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Patients With POAG or OHT
Number analyzed (Participants) | 315
mmHg | -4.2 (5.0)

ADVERSE EVENTS:
Arm/Group | Patients With POAG or OHT
Serious Adverse Events (participants affected / at risk) | 0/358
Other Adverse Events (participants affected / at risk) | 23/358
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With POAG or OHT (N=358)
Conjunctival hyperemia (Eye disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.